CLINICAL TRIAL: NCT01421108
Title: The Effectiveness of Gain- Versus Loss-framed Health Messages to Improve Oral Health Among Iranian Adolescents:A Randomized Controlled Trial
Brief Title: The Effectiveness of Gain- Versus Loss-framed Health Messages to Improve Oral Health Among Iranian Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qazvin University Of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir H Pakpour, Assistant professor, Qazvin University Of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACTRN12611000885998
Record Dates: First submitted 2011-08-12; First posted 2011-08-22 (Estimated); Last update posted 2012-03-06 (Estimated); Status verified 2012-03

CONDITIONS: Health Behavior
Keywords: oral health; dental brushing; dental flossing
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Loss-framed messages (Experimental)
  Interventions: Behavioral: Framing (Loss-framed messages)
- gain-framed messages (Experimental): Adolescents will randomly assign to three groups: gain-framed message , loss-framed message and a control group. Each group of adolescents will read the respective pamphlets with the exception of the control group. The gain-framed pamphlet contains six positive messages with three related full-color images (6.1 X 4.5). The gain-framed pamphlet, entitled The Benefits of good oral hygiene", emphasizes the benefits of brushing, and flossing.
  Interventions: Behavioral: Framing (Gain-framed messages)

INTERVENTIONS:
Behavioral: Framing (Gain-framed messages) — The adolescents will randomly assign to three groups: gain-framed message and loss- framed message. Each group of adolescents will read the respective pamphlets with the exception of the control group. The gain-framed pamphlet contains six positive messages with three related full-color images(6.1 X 4.5). The gain-framed pamphlet, entitled The Benefits of good oral hygiene", emphasizes the benefits of brushing, and flossing.
  Other Names: designing persuasive messages
  Arms: gain-framed messages
Behavioral: Framing (Loss-framed messages) — The adolescents will randomly assign to three groups: gain-framed message , loss- framed message and a control group. Each group of adolescents will read the respective pamphlets with the exception of the control group.
  The loss-framed pamphlet contains six negative messages with three related full-color images (6.1 X 4.5). The loss-framed pamphlet, entitled The disadvantages of poor oral hygiene, emphasizes the costs of not brushing and flossing.
  Arms: Loss-framed messages

SUMMARY:
This study explores the effectiveness of message framing, loss-framed vs. gain-framed messages on oral health in Iran.

DETAILED DESCRIPTION:
This is a study to explore the impact of two pamphlets with gain-framed and loss-framed messages on brushing and flossing attitudes, intentions , behaviors and clinical characteristics among a sample of adolescent students.

ELIGIBILITY:
Inclusion Criteria:

* They are not involved in the oral health education
* Ability to understand Persian language Adolescents attending high schools in Qazvin

Exclusion Criteria:

* Does not meet inclusion criteria

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 372 (Actual)
Dates: Start 2011-07; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
changes in frequencies of dental brushing and flossing | changes from baseline, two weeks after the intervention and six months follow-up

SECONDARY OUTCOMES:
Changes in psychological predictors of dental brushing (attitude, intention). | changes from baseline, two weeks after the intervention and six months follow-up
Changes in Community Periodontal Index (CPI) | changes from baseline, two weeks after the intervention and six months follow-up
Changes in Turesky Modification of the Quigley-Hein Plaque Index | changes from baseline, two weeks after the intervention and six months follow-up
Oral health related quality of life | changes from baseline and six months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Amir H Pakpour, PhD, Study Chair — Qazvin university medical of sciences
Locations (1):
- The Organization for Education, Qazvin, Qazvin Province, Iran

REFERENCES:
- [Derived] Pakpour AH, Yekaninejad MS, Sniehotta FF, Updegraff JA, Dombrowski SU. The effectiveness of gain-versus loss-framed health messages in improving oral health in Iranian secondary schools: a cluster-randomized controlled trial. Ann Behav Med. 2014 Jun;47(3):376-87. doi: 10.1007/s12160-013-9543-1. PMID 24163187